CLINICAL TRIAL: NCT04350775
Title: Investigation of Community Reablement on Instrumental Activities of Daily Living in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCHIRB-10812015
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia
Keywords: reablement; instrumental activities of daily living
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RE-IADL group (Experimental): Reablement
  Interventions: Other: RE-IADL
- Control group (Placebo Comparator): General community rehabilitation
  Interventions: Other: General community rehabilitation

INTERVENTIONS:
Other: RE-IADL — RE-IADL program is to conduct trainings related to instrumental activities of daily living. For example,using communication appliance, moving in community, financial management, health care, housework, prepare meals and clear ,and shopping.
  Arms: RE-IADL group
Other: General community rehabilitation — General community rehabilitation contains the activities in psychiatric rehabilitation center.
  Arms: Control group

SUMMARY:
This is a randomized controlled behavioral intervention trial to assess the efficacy of investigating program of Reablement-Instrumental Activities of Daily Living (RE-IADL) on schizophrenia patients at immediately and long-term.

DETAILED DESCRIPTION:
Subjects will be randomized to intervention group and control group. The outcome measures include the Canadian Occupational Performance Measure, Instrumental Activities of Daily Living-3 Dimensions, Activities of Daily Living Rating Scale III, Frenchay Activities Index, Lawton Instrumental Activities of Daily Living, Mini Mental State Examination-2nd edition, Behavior Rating Inventory of Executive Function adult version, Allen Cognitive Level Screen-6th, Participation Measure-3 Domains, 4 Dimensions, Personal and Social Performance scale, Work Behavior Inventory, Schizophrenia-Quality of Life questionnaire, Beck Depression Inventory-II, and Functioning Scale of the Disability Evaluation System.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by DSM-5
* age > 20 years
* Stable mental symptoms
* Willing to sign the subject's consent

Exclusion Criteria:

* History of severe brain injury
* Substance abuse
* Diagnosis of intellectual developmental disorder
* Unable to follow instructions

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Changes of the Canadian Occupational Performance Measure | 18 weeks
  The Canadian Occupational Performance Measure assesses occupational performance. A higher score indicates better occupational performance. Changes of the Canadian Occupational Performance Measure will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Instrumental Activities of Daily Living-3 Dimensions | 18 weeks
  The Instrumental Activities of Daily Living-3 Dimensions assesses instrumental activities of daily living about 3 Dimensions. A higher score indicates better instrumental activities of daily living. Changes of the Instrumental Activities of Daily Living-3 Dimensions will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Activities of Daily Living Rating Scale III | 18 weeks
  The Activities of Daily Living Rating Scale III assesses activities of daily living. A higher score indicates better activities of daily living. Changes of the Activities of Daily Living Rating Scale III well be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Frenchay Activity Index | 18 weeks
  The Frenchay Activity Index assesses instrumental activities of daily. A higher score indicates better instrumental activities of daily living. Changes of the Frenchay Activity Index will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Lawton Instrumental Activities of Daily Living | 18 weeks
  The Lawton Instrumental Activities of Daily Living assesses instrumental activities of daily living. A higher scores indicates better instrumental activities of daily living. Changes of the Lawton Instrumental Activities of Daily Living will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Mini Mental State Examination-2nd edition | 18 weeks
  The Mini Mental State Examination assesses general cognitive function. A higher score indicates better general cognitive function. Changes of the Mini Mental State Examination will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Behavior Rating Inventory of Executive Function adult version | 18 weeks
  The Behavior Rating Inventory of Executive Function adult version assesses executive functions. A lower score indicates better executive functions. Changes of the Behavior Rating Inventory of Executive Function adult version will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Allen Cognitive Level Screen-6th | 18 weeks
  The Allen Cognitive Level Screen-6th assesses cognitive functions. A higher score indicates better cognitive functions. Changes of the Allen Cognitive Level Screen-6th will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Participation Measure-3 Domains, 4 Dimensions | 18 weeks
  The Participation Measure-3 Domains, 4 Dimensions assesses social participation. A higher score indicates better social participation. Changes of the Participation Measure-3 Domains, 4 Dimensions will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Personal and Social Performance scale | 18 weeks
  The Personal and Social Performance scale assesses social functioning. A higher score indicates better social functioning. Changes of the Personal and Social Performance scale will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Work Behavior Inventory | 18 weeks
  The Work Behavior Inventory assesses work behavior about chronic mental patients. A lower score indicates better work behavior. Changes of the Work Behavior Inventory will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Schizophrenia-Quality of Life questionnaire | 18 weeks
  The Schizophrenia-Quality of Life questionnaire assesses schizophrenia quality of life. A higher score indicates better quality of life. Changes of the Schizophrenia-Quality of Life questionnaire will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Beck Depression Inventory-II | 18 weeks
  The Beck Depression Inventory-II assesses the person about depression. A higher score indicates more depression. Changes of the Beck Depression Inventory-II will be assessed at the 0 week, 6 weeks, and 18 weeks.
Changes of the Functioning Scale of the Disability Evaluation System | 18 weeks
  The Functioning Scale of the Disability Evaluation System assesses status of individuals' activities and participation. A higher score indicates more barriers or limitations. Changes of the Functioning Scale of the Disability Evaluation System will be assessed at the 0 week, 6 weeks, and 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Wanhua Dist, Taiwan